CLINICAL TRIAL: NCT02445443
Title: A Prospective, Multi-center Clinical Study Evaluating the LEGION™ Hinge Knee System
Brief Title: LEGION Hinge Safety and Efficacy Study
Acronym: LINKS
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-4042-01
Record Dates: First submitted 2015-04-30; First posted 2015-05-15 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LEGION Hinge Knee System: This group will be receiving the LEGION Hinge device.
  Interventions: Device: LEGION Hinge Knee System

INTERVENTIONS:
Device: LEGION Hinge Knee System — All enrolled/treated subjects will receive the LEGION Hinge Knee System.
  Other Names: LEGION HK

SUMMARY:
The purpose of the current investigation is to assess the safety and efficacy of a new hinged revision knee device. This device is designed to provide efficient, reproducible reconstructions with optimal limb and implant alignment, durable implant fixation, and functional outcomes that increasingly approach those of primary Total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
The objective of this study is to demonstrate statistically significant improvements in the original Knee Society Clinical Score (KSCS) from baseline to 1 and 2 years in subjects using the LEGION™ Hinge Knee System. The focus of the 1 and 2 year analyses will be on safety and efficacy. The 5 year analysis will focus on survivorship and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject has gross knee instability resulting from loss of collateral ligament function, gross bone loss, comminuted fractures of the proximal tibia or distal femur, rheumatoid arthritis, post-traumatic arthritis, osteoarthritis, degenerative arthritis, failed osteotomies, unicompartmental replacement or total knee replacement, or absent or incompetent posterior cruciate ligament and one or both of the collateral ligaments
* Subject has a failed primary or revision knee replacement
* Subject is 18-80 years of age
* Subject is skeletally mature in Investigator's judgment i.e., subject is not actively growing or does not have immature bones for any reason
* Subject has met an acceptable preoperative medical clearance and is free of or treated for cardiac, pulmonary, hematological, infection or other conditions that would pose excessive operative risk
* Subject is willing to sign and date an IRB/EC-approved consent form
* Subject plans to be available through the five (5) year postoperative follow-up
* If of child bearing potential, Subject reports she is not pregnant nor plans to become pregnant during the study
* Subject agrees to follow the study protocol

Exclusion Criteria:

* Subject is receiving the study device as a primary knee replacement
* Subject has presence of malignant tumor, metastatic, or neoplastic disease
* Subject is not expected to return to normal ambulatory function (i.e., morbid obesity or other limiting co-morbidities)
* Subject is pregnant or plans to become pregnant during the course of the study
* Subject has conditions that may interfere with the revision arthroplasty survival or outcome (i.e., Paget's or Charcot-Marie-Tooth disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease)
* Subject has known (Subject reported) metal hypersensitivity
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in this study
* Subject has BMI>45
* Subject is participating in any other pharmaceutical, biologic, or medical device clinical investigation or has been treated with an investigational product in the past 30 days
* Subject is facing current or impending incarceration
* Subject is not a good candidate for the study based on Investigator opinion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a revision total knee arthroplasty (TKA) using the LEGION Hinge Total Knee system.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Original Knee Society Clinical Score© (KSCS) | 1 year
  The original Knee Society Score© (KSS) is subdivided into two parts. One part is the Knee Society Clinical Score (KSCS) and the other part is the Knee Society Functional Score (KSFS). The KSCS will be administered at the pre-operative visit and all follow-up visits. The purpose of administering this assessment is to determine the statistical clinical improvement over time which may be compared to literature at 1 and 2 years.
Revision | Up to 5 years
  Revision, for any reason, will be assessed throughout the subject's participation in the study.

SECONDARY OUTCOMES:
Original Knee Society Functional Score© (KSFS) | 1 year
  The original Knee Society Score© (KSS) is subdivided into two parts. One part is the Knee Society Clinical Score (KSCS) and the other part is the Knee Society Functional Score (KSFS). The purpose of administering this assessment is to determine the statistical clinical improvement over time which may be compared to literature at 1 and 2 years.
Original Knee Society Functional Score© (KSFS) | 2 years
  The original Knee Society Score© (KSS) is subdivided into two parts. One part is the Knee Society Clinical Score (KSCS) and the other part is the Knee Society Functional Score (KSFS). The purpose of administering this assessment is to determine the statistical clinical improvement over time which may be compared to literature at 1 and 2 years.
2011 Knee Society Score© | 1 year
  2011 Knee Society Knee Score and all of it's components
2011 Knee Society Score© | 2 years
  2011 Knee Society Knee Score and all of it's components
EQ-5D-3L™ | 1 year
  The EuroQol EQ-5D-3L™ is a descriptive system measuring health-related Quality Of Life (QOL) and consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D-3L™ dimension. The EQ-5D-3L™ is completed by the Subject on the day of their visit.
EQ-5D-3L™ | 2 years
  The EuroQol EQ-5D-3L™ is a descriptive system measuring health-related Quality Of Life (QOL) and consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which takes one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D-3L™ dimension. The EQ-5D-3L™ is completed by the Subject on the day of their visit.
Original Knee Society Clinical Score© (KSCS) | 2 Years
  The original Knee Society Score© (KSS) is subdivided into two parts. One part is the Knee Society Clinical Score (KSCS) and the other part is the Knee Society Functional Score (KSFS). The KSCS will be administered at the pre-operative visit and all follow-up visits. The purpose of administering this assessment is to determine the statistical clinical improvement over time which may be compared to literature at 1 and 2 years.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - University of Iowa Hospitals, Iowa City, Iowa
  - NYU Hospital for Joint Diseases, New York, New York
  - Oregon Health and Science University, Portland, Oregon
- Fremantle Hospital, Fremantle, Western Australia, Australia
- UZ Leuven campus Pellenberg, Pellenberg, Belgium
- Concordia Hip and Knee Institute, Winnipeg, Manitoba, Canada
- University Hospital Mutua de Terrassa, Terrassa, Barcelona, Spain